CLINICAL TRIAL: NCT03978429
Title: A Cluster Randomized, Parallel-group, Superiority Study to Compare the Effectiveness of a Community-based mHealth Strategy Versus Enhanced Usual Care in the Detection and Management of Pre-eclampsia/Eclampsia in Tanzania
Brief Title: An mHealth Strategy to Reduce Pre-Eclampsia and Infant Death in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Karen Yeates (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. Karen Yeates, Professor, Department of Medicince, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 108022
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced
Keywords: Pre-eclampsia; Eclampsia; mHealth; mobile health; Gestosis; Hypertension, Pregnancy-Induced
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and health providers in the control clinics are unaware of the intervention and the investigators and outcome assessors are completely blinded from assignment of the intervention to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): 1. Community-based Pre-eclampsia/Eclampsia Detection and Management
  2. Strengthened Referral Network from Community to Referral hospital levels
  3. Antenatal Care Nurses will receive training on best practices for PE detection and management per Tanzanian Standard Treatment Guidelines.
  4. Antenatal Care Nurses will be given smartphones and will be trained to complete Case Report Forms (CRF) to log key indicators and activities at each ANC visit, delivery and Postnatal Care visits of enrolled participants.
  5. Antenatal Care Nurses will receive bluetooth blood pressure monitors.
  6. Community Health Workers within the intervention arm facilities will receive training in pre-eclampsia features and will be provided with smart phones and access to a smart phone application that will prompt them to initiate follow ups with pregnant women within the community and they will receive SMS/text messages reminders about pregnant women within the community who require follow up.
  Interventions: Other: Community-based Pre-eclampsia/Eclampsia Detection and Management; Other: Strengthened Referral Network from Community to Referral hospital levels
- Enhanced Usual Care (No Intervention): 1. Antenatal Care Nurses will receive training on best practices for PE detection and management per Tanzanian Standard Treatment Guidelines.
  2. Antenatal Care Nurses will be given smartphones and will be trained to complete Case Report Forms (CRF) to log key indicators and activities at each ANC visit, delivery and Postnatal Care visits of enrolled participants.
  3. Antenatal Care Nurses will receive bluetooth blood pressure monitors.

INTERVENTIONS:
Other: Community-based Pre-eclampsia/Eclampsia Detection and Management — Three Community Health Workers (CHWs) per health facility (cluster) will be equipped with android smartphones and blood pressure monitors. The CHWs will visit participant's home once per month until 6 weeks post-partum and complete a Case Report Form for signs and symptoms of pre-eclampsia and blood pressure. CHWs, Antenatal Care Nurses (ANC) at the woman's health facility and study coordinator will receive SMS message if the algorithm on our platform (informed by the Tanzanian Standard Treatment Guidelines (TSTG) deems she is at risk for pre-eclampsia. This message will indicate that the woman needs to be referred to her health facility if: participant has high blood pressure, a significant intrapatient rise in blood pressure or a combination of factors according to an algorithm. Woman's condition will be assessed and ANC will decide on the management, including rest at home with CHW monitoring. Women found to be at risk for pre-eclampsia will be visited twice monthly.
  Arms: Intervention Arm
Other: Strengthened Referral Network from Community to Referral hospital levels — ANC nurses and CHWs will play complementary roles in performing activities to meet key indicators and facilitate referrals. They will deliver a plan using the Pre-eclampsia application tool on their smart phone and then they can refer the pregnant woman for enrollment for facility care and track them as per key indicators. The key innovation is that the mHealth platform can detect increases in BP within each patient, and this ability to detect is brought down to the community level through CHWs. This will allow for earlier detection of PE as singular BPs. Nurses will receive protocolized instructions and education regarding when to refer a woman to a higher-level facility for further management. The program consists of SMS component delivered to provide information about participant's condition to relevant members of the referral pathway to enhance referrals and facilitate community level follow up.
  Arms: Intervention Arm

SUMMARY:
The core of this study is a cluster randomized controlled trial (RCT) of antenatal clinics which are located in four districts in Tanzania. We are conducting an effectiveness (pragmatic) rather than an efficacy (explanatory) trial because we are looking to measure the degree of benefit under 'real world' conditions. Although pragmatic and carried out in real world conditions, the proposed size and scope of the trial will allow us to achieve a robust evaluation of outcomes and determine the effectiveness of our intervention. A cluster design is the most appropriate type of methodology (rather than individual randomization by pregnant woman) as the intervention can be delivered to the entire health facility (of those facilities in the intervention group). The intervention is to implement an mHealth strategy to improve detection and management of PE (pre-eclampsia). This study is a multi-level, mixed-methods design that includes a cluster-randomized controlled trial (RCT) of antenatal clinics in rural Tanzania. Thirty health facilities have been randomized to control facilities and thirty facilities have been randomized to intervention clinics. All randomized clinics have upgraded antenatal care (ANC) and skilled birth attendants present. Nurses in the intervention clinics in this cluster arm will receive mHealth-based education in detection and management of PE and will be instructed and encouraged to follow a guideline-driven approach supported by mHealth (educational modules that provide decision support and reminders through the facility smartphone/tablet). At all antenatal visits, pregnant women will have their blood pressures measured and urine assessed for proteinuria, and, the result will be automatically sent by SMS (short message service) with a unique patient identifier to a central site for monitoring and tracking. Community Health Workers (CHWs) linked to the facility site and local communities will be instructed on which women to have follow-up visits within their communities. For all those women found to be at risk for PE (as well as other high risk maternal conditions), an SMS will be sent to the CHW, and, the nurses at the ANC recommending timely follow-up and protocol steps for management at that facility or for transfer for further monitoring and management at a higher-level facility. The nurses participating in the study have been drawn from the health facilities themselves, in both control and intervention arms. Quantitative data will be collected on an ongoing basis through the mobile platform. Women are eligible for recruitment between 15 weeks and 36 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* at least 5 months pregnant

Exclusion Criteria:

* Unable to provide consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 3000 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome (composite indicator reflecting activities associated with recognition and management/treatment of pre-eclampsia) | Outcome is evaluated at one month post delivery
  A composite indicator reflecting activities (1) associated with recognition of pre-eclampsia by recognizing 1 of these 4 items; Blood pressure reading greater than 140 mmHg, Diastolic greater than 90 mmHg, Intrapatient BP rise of 30mmHg systolic or 15mmHg diastolic, Proteinuria (+) and headache, visual disturbance or both and/or epigastric pain and vomiting, or both, or edema and (2)activities associated with the management/treatment of pre-eclampsia.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Yeates, MD, Principal Investigator — Queen's University
Locations (1):
- Ifakara Health Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Bureau of Statistics,. Tanzania Demographic and Health Survey (TDHS-MIS) 2010. (MoHCDGEC, MoH, NBS, OCGS, and ICF, 2010).
- [Background] Ministry of Health, Community Development, Gender, Elderly and Children (MoHCDGEC) [Tanzania, Mainland], Ministry of Health (MoH) [Zanzibar], National Bureau of Statistics (NBS), Office of the Chief & Government Statistician (OCGS), and ICF. Tanzania Demographic and Health Survey and Malaria Indicator Survey (TDHS-MIS) 2015-16. (MoHCDGEC, MoH, NBS, OCGS, and ICF, 2016).
- [Background] The National Republic of Tanzania Ministry of Health, Community Development, Gender, Elderly and Children. Standard Treatment Guidelines & National Essential Medicines List. Fifth Edition. (2017).
- [Background] Maar MA, Yeates K, Toth Z, Barron M, Boesch L, Hua-Stewart D, Liu P, Perkins N, Sleeth J, Wabano MJ, Williamson P, Tobe SW. Unpacking the Black Box: A Formative Research Approach to the Development of Theory-Driven, Evidence-Based, and Culturally Safe Text Messages in Mobile Health Interventions. JMIR Mhealth Uhealth. 2016 Jan 22;4(1):e10. doi: 10.2196/mhealth.4994. PMID 26800712
- [Background] Rosenstock, I. M. The Health Belief Model and Preventive Health Behavior. Health Educ. Behav. 2, 354-386 (1974).
- [Background] Jennings L, Gagliardi L. Influence of mHealth interventions on gender relations in developing countries: a systematic literature review. Int J Equity Health. 2013 Oct 16;12:85. doi: 10.1186/1475-9276-12-85. PMID 24131553
- [Background] Research in Gender and Ethics (RinGs). mHealth and Gender: Making the Connection. (2015).
- [Background] Nie J, Unger JA, Thompson S, Hofstee M, Gu J, Mercer MA. Does mobile phone ownership predict better utilization of maternal and newborn health services? a cross-sectional study in Timor-Leste. BMC Pregnancy Childbirth. 2016 Jul 23;16(1):183. doi: 10.1186/s12884-016-0981-1. PMID 27448798
- [Background] GSMA Intelligence. Bridging the gender gap: Mobile access and usage in low- and middle-income countries. (2016).
- [Background] GSMA Intelligence. Women and Mobile: A Global Opportunity.
- [Background] Wesolowski A, Eagle N, Noor AM, Snow RW, Buckee CO. Heterogeneous mobile phone ownership and usage patterns in Kenya. PLoS One. 2012;7(4):e35319. doi: 10.1371/journal.pone.0035319. Epub 2012 Apr 25. PMID 22558140
- [Background] Blumenstock, J. & Eagle, N. Mobile divides: gender, socioeconomic status, and mobile phone use in Rwanda. in Proceedings of the 4th ACM/IEEE International Conference on Information and Communication Technologies and Development 6 (ACM, 2010).
- [Background] GSMA mWomen. Striving and Surviving: Exploring the Lives of Women at the Base of the Pyramid. 1-74 (2012).
- [Background] Chib A, Wilkin H, Ling LX, Hoefman B, Van Biejma H. You have an important message! Evaluating the effectiveness of a text message HIV/AIDS campaign in Northwest Uganda. J Health Commun. 2012;17 Suppl 1:146-57. doi: 10.1080/10810730.2011.649104. PMID 22548607
- [Background] Siedner MJ, Santorino D, Haberer JE, Bangsberg DR. Know your audience: predictors of success for a patient-centered texting app to augment linkage to HIV care in rural Uganda. J Med Internet Res. 2015 Mar 24;17(3):e78. doi: 10.2196/jmir.3859. PMID 25831269
- [Background] Eichler M, Burke MA. The BIAS FREE Framework: a new analytical tool for global health research. Can J Public Health. 2006 Jan-Feb;97(1):63-8. doi: 10.1007/BF03405218. PMID 16512332
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394